CLINICAL TRIAL: NCT00214968
Title: A 6-Month Open Label, Flexible-Dosage Study to Assess the Safety and Effectiveness of PROVIGIL (Modafinil) Treatment in Children and Adolescents With Excessive Sleepiness Associated With Narcolepsy or Obstructive Sleep Apnea/Hypopnea Syndrome
Brief Title: Assess the Safety and Effectiveness of PROVIGIL Treatment in Children and Adolescents With Excessive Sleepiness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1538/3034/ES/MN
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Narcolepsy
MeSH Terms: conditions — Narcolepsy | interventions — Modafinil

ARMS (1):
- Modafinil (Experimental): Subjects began taking Provigil at a dosage of 100 mg/day (1 tablet) and increased their dosage by 100 mg/day each week for up to 4 weeks
  Interventions: Drug: Modafinil

INTERVENTIONS:
Drug: Modafinil — maximum dosage 400 mg/day (4 tablets)
  Other Names: Provigil

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of treatment with PROVIGIL in children and adolescents with excessive sleepiness (ES) associated with narcolepsy or obstructive sleep apnea/hypopnea syndrome (OSAHS), when administered for up to 6 months.

ELIGIBILITY:
Inclusions Criteria:

* written informed consent/assent is obtained
* meet minimal criteria established by the International Classification of Sleep Disorders (ICSD) manual of the American Academy of Sleep Medicine (AASM) for narcolepsy (or presumed narcolepsy) or OSAHS OR have a previous diagnosis of narcolepsy or OSAHS before the screening visit
* have a complaint of ES
* are in good health as determined by a medical and psychiatric history, physical examination, ECG, and clinical laboratory tests
* have blood pressure values greater than those for the 5th percentile and less than the 95th percentile on the National High Blood Pressure Education Program guidelines for blood pressure levels for boys and girls ages 6 to 16 years
* girls who are postmenarchal or sexually active, have a negative urine pregnancy test at screening, must be using a medically acceptable method of birth control, and must agree to continue use of this method for the duration of the study (and for 2 cycles after participation in the study); acceptable methods of birth control include: barrier method with spermicide; steroidal contraceptives (oral, transdermal, implanted, or injected) in conjunction with a barrier method; intrauterine device (IUD); or abstinence
* able to swallow a tablet similar in size and shape to the study drug tablet
* negative urine drug screen (UDS) for any illicit drug, alcohol (ethanol), stimulants at screening; if positive for stimulants (prescribed for excessive sleepiness) at screening, UDS to be repeated after a washout period and before baseline
* have a parent or legal representative who is willing to participate in the study

Exclusion Criteria:

* have self-induced sleep deprivation/poor sleep hygiene
* have a past or present seizure disorder (except history of single febrile seizure), a history of psychosis, or of clinically significant head trauma (eg, brain damage) or past neurosurgery
* have a history of suicide attempt, or are at suicidal risk
* a clinically significant drug sensitivity to stimulants such as amfetamine, dexamfetamine, or methylphenidate; and/or modafinil or any of its components
* use of any monoamine oxidase (MAO) inhibitors or selective serotonin reuptake inhibitors (SSRIs) within 2 weeks of the baseline visit (NOTE: SSRIs will be allowed for cataplexy if the patient has been on a stable dose for at least 1 month.)
* received any investigational drug (except modafinil) within 4 weeks of the baseline visit
* any disorder that could interfere with drug absorption, distribution, metabolism, or excretion (including previous gastrointestinal surgery)
* active, clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematologic, neoplastic, endocrine, neurologic, immunodeficiency, pulmonary, or other major clinically significant disorder/disease
* any clinically significant deviation from the normal range(s) in the physical examination or ECG findings, or clinical laboratory test results (ie, serum chemistry, hematology) at the screening or baseline visit
* absolute neutrophil count (ANC) below the lower limit of normal at screening (NOTE: If the ANC is below the lower limit of normal at the baseline visit, the medical monitor will be consulted for continued eligibility in the study.)
* a history of alcohol, narcotic, or any other substance abuse
* pregnant or lactating/nursing girl

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2005-01; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Adverse event evaluations | up to 6 months
  Evaluate the safety and tolerability of treatment in children and adolescents with excessive daytime sleepiness associated with narcolepsy and obstructive sleep apnea/hypopnea syndrome, when administered for up to 6 months

SECONDARY OUTCOMES:
Composite Ratings of severity of illness | up to 6 months
  Clinical global impression (CGI-C) ratings for severity of illness. The ratings range from 1 to 7; 1 =normal-not at all ill to 7 =among the most extremely ill.
Total score from the Pediatric Daytime Sleepiness Scale (PDSS) | up to 6 months
  A measure of daytime sleepiness and school-related outcomes using PDSS questions: This self-report 8-item questionnaire asks questions with ranges from Always to Never; always being the worst case and never the best case.